CLINICAL TRIAL: NCT00171730
Title: Extension to a Multi-Center, Randomized, Crossover, Open Label, Dose Finding Study to Compare the Safety, Efficacy, and Pharmacokinetics/Pharmacodynamics (PK/PD) Relationship of Multiple Doses of Pasireotide (SOM230) (200, 400, and 600 μg Bid) and Doses of Open Label Sandostatin® (SMS) (100 μg Tid) in Acromegalic Patients
Brief Title: An Extension Study to Assess the Long-Term Safety and Efficacy of Pasireotide in Participants With Acromegaly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2201E1; 2004-002849-12 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Acromegaly
Keywords: Acromegaly; Pasireotide; GH; IGF-1
MeSH Terms: conditions — Acromegaly | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pasireotide s.c. Overall (Experimental): Participants received pasireotide as a daily subcutaneous (s.c) injection, every 12 hours at 9:00 AM and 9:00 PM at the dose at which the biochemical control was achieved (either 200, 400, or 600 microgram (μg)) for as long as the participant benefited from the treatment, and there were no safety or tolerability concerns (median duration of 22.7 months).
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide
  Other Names: SOM230

SUMMARY:
Acromegaly is a rare, serious condition characterized by chronic hypersecretion of growth hormone (GH), generally caused by a GH-secreting pituitary adenoma. The study assessed the long-term safety and efficacy of pasireotide in participants with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed all four treatment regimens in the core study CSOM230B2201 (NCT00088582) and achieved biochemical control in growth hormone (GH) and insulin-like growth factor-1 (IGF-1) levels after at least one month of pasireotide administration at any of the three doses.
* Participants who did not experience any unacceptable adverse events or tolerability issues during the core study CSOM230B2201.

Exclusion Criteria:

* Participants who experienced or developed compression of the optic chiasm causing any visual field defect during the core study CSOM230B2201.
* Participants who required a surgical intervention for relief of any sign or symptom associated with tumor compression during the core study CSOM230B2201.
* Participants who experienced or developed congestive heart failure, unstable angina, sustained ventricular tachycardia, ventricular fibrillation or acute myocardial infraction during the core study CSOM230B2201.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-08-24 (Actual); Primary Completion 2013-12-06 (Actual); Study Completion 2013-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (10):
- United States (3):
  - Cedars Sinai Medical Center Dept. of Pituitary Ctr., Los Angeles, California
  - University of Michigan Health System StudyCoordinatorCSOM230B2201E1, Ann Arbor, Michigan
  - NYU / VA Medical Center, New York, New York
- Novartis Investigative Site, Woolloongabba, Queensland, Australia
- Novartis Investigative Site, Edegem, Belgium
- Novartis Investigative Site, Toulouse Cédex 4, France
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Novartis Investigative Site, Napoli, Italy
- Novartis Investigative Site, Lausanne, Switzerland

REFERENCES:
- [Result] Petersenn S, Farrall AJ, De Block C, Melmed S, Schopohl J, Caron P, Cuneo R, Kleinberg D, Colao A, Ruffin M, Hermosillo Resendiz K, Hughes G, Hu K, Barkan A. Long-term efficacy and safety of subcutaneous pasireotide in acromegaly: results from an open-ended, multicenter, Phase II extension study. Pituitary. 2014 Apr;17(2):132-40. doi: 10.1007/s11102-013-0478-0. PMID 23529827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study was an open label, single arm, multi-center study in participants with acromegaly who had completed all four treatment regimens in the core study CSOM230B2201 (NCT00088582) and achieved biochemical control or had clinically relevant improvement according to Investigator judgement, from at least one of the pasireotide regimens.
Pre-assignment Details: Baseline visit in this extension study is referred as Month 3 which was the end of core study. Subsequent visits occurred at every 3 months (referred as Months 6, 9, 12 and so on) till the end of this study.
Groups:
- Pasireotide s.c. Overall: Participants received pasireotide as a daily subcutaneous (s.c.) injection every 12 hours at 9:00 AM and 9:00 PM at the dose at which the biochemical control was achieved (either 200, 400, or 600 μg) for as long as the participant benefited from the treatment, and there were no safety or tolerability concerns (median duration of 22.7 months).
Period: Overall Study
Arm/Group | Pasireotide s.c. Overall
Started | 30
Completed | 15
Not Completed | 15
Not completed — Adverse Event | 3
Not completed — Abnormal Laboratory Value(s) | 1
Not completed — Unsatisfactory Therapeutic Effect | 8
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received pasireotide s.c. in the extension study.
Groups:
- Pasireotide s.c. Overall: Participants received pasireotide as a daily s.c. injection every 12 hours at 9:00 AM and 9:00 PM at the dose at which the biochemical control was achieved (either 200, 400, or 600 μg) for as long as the participant benefited from the treatment, and there were no safety or tolerability concerns (median duration of 22.7 months).
Arm/Group | Pasireotide s.c. Overall
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Growth Hormone (GH) and Insulin-like Growth Factor 1 (IGF-1) Observed Response by Dose Class
Description: A participant was a responder to a dose level if the mean GH level after dosing (t30, t60, t90, and t120) was below/equal to 2.5 microgram/litre (μg/L), and if the mean of IGF-1 of the two pre-dose values (t-30, t-1) was within normal limits for age-sex matched controls. If three or more of t30, t60, t90, or t120 were missing, mean GH was considered missing. If either t-30 or t-1 was missing, mean IGF-1 was considered missing. Pasireotide incident dose classes were defined by total daily doses ranges (<1200 μg/d, 1200 to <1500 μg/d, ≥ 1500 μg/d).
Time Frame: Month 9 (Month 9 visit is at the completion of six months in this extension study)
Population: Efficacy analyzable population included all participants who received at least one dose of pasireotide during the extension study and had at least one post-extension baseline efficacy evaluation. Overall number of participants analyzed is the number of participants with at least 2 GH measurements and both predose IGF-1 measurements at the corresponding visit.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- Pasireotide s.c. <1200 μg/d: Participants received pasireotide as a daily s.c. injection every 12 hours at 9:00 AM and 9:00 PM at the dose at which the biochemical control was achieved (either 200, 400, or 600 μg), with total daily dose <1200 μg/day with median duration of 2.1 months.
- Pasireotide s.c. 1200 to <1500 μg/d: Participants received pasireotide as a daily s.c. injection every 12 hours at 9:00 AM and 9:00 PM at the dose at which the biochemical control was achieved (either 200, 400, or 600 μg), with total daily dose 1200 to <1500 μg/day with median duration of 6.4 months.
- Pasireotide s.c. ≥1500 μg/d: Participants received pasireotide as a daily s.c. injection every 12 hours at 9:00 AM and 9:00 PM at the dose at which the biochemical control was achieved (either 200, 400, or 600 μg), with total daily dose ≥ 1500 μg/day with median duration of 16.6 months.
Arm/Group | Pasireotide s.c. <1200 μg/d | Pasireotide s.c. 1200 to <1500 μg/d | Pasireotide s.c. ≥1500 μg/d | Pasireotide s.c. Overall
Number analyzed (Participants) | 5 | 14 | 7 | 26
percentage of responders | 20 [9.0 to 43.6] | 28.6 [9.0 to 43.6] | 14.3 [9.0 to 43.6] | 23.1 [9.0 to 43.6]

2. Secondary Outcome: Time to Tumor Response
Description: Time to tumor response was defined as time from Sandostatin baseline (core study baseline) to at least 20% decrease in tumor volume.
Time Frame: Core study baseline to at least a 20% decrease in pituitary tumor volume (up to approximately 114 months)
Population: Efficacy analyzable population included all participants who received at least one dose of pasireotide during the extension study and had at least one post-extension baseline efficacy evaluation. Overall number of participants analyzed is the number of participants with data available at the specified time point.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pasireotide s.c. Overall
Number analyzed (Participants) | 29
months | 12.2 [4.9 to 19.2]

3. Secondary Outcome: Summary Magnetic Resonance Imaging (MRI) Pituitary Tumor Volumes
Description: Pituitary Tumor Volumes were assessed by MRI. Core study baseline was defined as the last non-missing observation prior to the start of Sandostatin s.c. treatment.
Time Frame: Core study baseline, Months 9, 27, 63, 75 and 99
Population: Efficacy analyzable population included all participants who received at least one dose of pasireotide during the extension study and had at least one post-extension baseline efficacy evaluation. Number analyzed is the number of participants with data available at specified time points.
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm)
Arm/Group | Pasireotide s.c. Overall
Number analyzed (Participants) | 30
cubic millimeter (mm)
  Core Study Baseline: number analyzed (Participants) | 29
  Core Study Baseline | 4457.4 (4891.98)
  Month 9: number analyzed (Participants) | 16
  Month 9 | 2839.3 (2710.61)
  Month 27: number analyzed (Participants) | 5
  Month 27 | 2536 (2219.13)
  Month 63: number analyzed (Participants) | 2
  Month 63 | 456 (381.84)
  Month 75: number analyzed (Participants) | 3
  Month 75 | 1016 (872.39)
  Month 99: number analyzed (Participants) | 1
  Month 99 | 180 (NA) — Due to one participant available for analysis standard deviation (SD) was not estimable.

4. Secondary Outcome: Percentage of Participants With Symptoms of Acromegaly
Description: Participants scored the following symptoms of acromegaly: Headache, perspiration, paresthesia, fatigue, osteoarthralgia, and carpal tunnel syndrome on a 5-point scale (0 = None/absent, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Very severe).
Time Frame: Core study baseline till the last assessment of the extension study (up to approximately 114 months)
Population: Efficacy analyzable population included all participants who received at least one dose of pasireotide during the extension study and had at least one post-extension baseline efficacy evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Pasireotide s.c. Overall
Number analyzed (Participants) | 30
percentage of participants
  Headache - 0 | 46.7
  Headache - 1 | 26.7
  Headache - 2 | 6.7
  Headache - 3 | 0
  Headache - 4 | 0
  Headache - Not Done | 20
  Perspiration - 0 | 20
  Perspiration - 1 | 33.3
  Perspiration - 2 | 23.3
  Perspiration - 3 | 3.3
  Perspiration - 4 | 0
  Perspiration - Not Done | 20
  Paresthesiae - 0 | 50
  Paresthesiae - 1 | 16.7
  Paresthesiae - 2 | 13.3
  Paresthesiae - 3 | 0
  Paresthesiae - 4 | 0
  Paresthesiae - Not Done | 20
  Fatigue - 0 | 26.7
  Fatigue - 1 | 26.7
  Fatigue - 2 | 13.3
  Fatigue - 3 | 13.3
  Fatigue - 4 | 0
  Fatigue - Not Done | 20
  Osteoarthralgia - 0 | 40
  Osteoarthralgia - 1 | 23.3
  Osteoarthralgia - 2 | 10
  Osteoarthralgia - 3 | 3.3
  Osteoarthralgia - 4 | 3.3
  Osteoarthralgia - Not Done | 20
  Carpal Tunnel Syndrome - 0 | 56.7
  Carpal Tunnel Syndrome - 1 | 10
  Carpal Tunnel Syndrome - 2 | 10
  Carpal Tunnel Syndrome - 3 | 3.3
  Carpal Tunnel Syndrome - 4 | 0
  Carpal Tunnel Syndrome - Not Done | 20

5. Secondary Outcome: Percentage of Participants With Sleep Apnea Symptoms as Assessed by Epworth Sleepiness Scale by Situation
Description: Sleep apnea symptoms were assessed using the Epworth Sleepiness Scale (ESS). The ESS is a self-administered questionnaire with 8 questions. It provides a measure of a person's general level of daytime sleepiness, or average sleep propensity in daily life. Percentage of participants were reported in 8 different situations: sitting and reading; watching TV; sitting, inactive in a public place; passenger in a car, an hour without break; lying down to rest in the afternoon; sitting and talking to someone; sitting quietly after a lunch without alcohol; and in a car, stopped a few minutes in the traffic. The participants were rated: 0 = would never doze, 1 = slight chance of dozing, 2 = moderate chance of dozing, 3 = high chance of dozing. Higher scores indicate more severe daytime sleepiness.
Time Frame: Core study baseline till the last assessment of the extension study (up to approximately 114 months)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pasireotide s.c. Overall
Number analyzed (Participants) | 30
percentage of participants
  Sitting and Reading - 0 | 36.7
  Sitting and Reading - 1 | 23.3
  Sitting and Reading - 2 | 23.3
  Sitting and Reading - 3 | 0
  Sitting and Reading - Not Done | 16.7
  Watching TV - 0 | 23.3
  Watching TV - 1 | 33.3
  Watching TV - 2 | 23.3
  Watching TV - 3 | 3.3
  Watching TV - Not Done | 16.7
  Sitting, Inactive in a Public Place - 0 | 56.7
  Sitting, Inactive in a Public Place - 1 | 20
  Sitting, Inactive in a Public Place - 2 | 6.7
  Sitting, Inactive in a Public Place - 3 | 0
  Sitting, Inactive in a Public Place - Not Done | 16.7
  Passenger in a Car, an Hour Without Break - 0 | 60
  Passenger in a Car, an Hour Without Break - 1 | 10
  Passenger in a Car, an Hour Without Break - 2 | 6.7
  Passenger in a Car, an Hour Without Break - 3 | 6.7
  Passenger in a Car, an Hour Without Break - Not Done | 16.7
  Lying Down to Rest in the Afternoon - 0 | 13.3
  Lying Down to Rest in the Afternoon - 1 | 23.3
  Lying Down to Rest in the Afternoon - 2 | 23.3
  Lying Down to Rest in the Afternoon - 3 | 23.3
  Lying Down to Rest in the Afternoon - Not Done | 16.7
  Sitting and Talking to Someone - 0 | 76.7
  Sitting and Talking to Someone - 1 | 6.7
  Sitting and Talking to Someone - 2 | 0
  Sitting and Talking to Someone - 3 | 0
  Sitting and Talking to Someone - Not Done | 16.7
  Sitting Quietly After a Lunch Without Alcohol - 0 | 30
  Sitting Quietly After a Lunch Without Alcohol - 1 | 23.3
  Sitting Quietly After a Lunch Without Alcohol - 2 | 20
  Sitting Quietly After a Lunch Without Alcohol - 3 | 10
  Sitting Quietly After a Lunch Without Alcohol - Not Done | 16.7
  In a Car, Stopped a Few Minutes in the Traffic - 0 | 73.3
  In a Car, Stopped a Few Minutes in the Traffic - 1 | 10
  In a Car, Stopped a Few Minutes in the Traffic - 2 | 0
  In a Car, Stopped a Few Minutes in the Traffic - 3 | 0
  In a Car, Stopped a Few Minutes in the Traffic - Not Done | 16.7

6. Secondary Outcome: Percentage of Participants With One or More Adverse Events (AEs)
Description: An AE was any undesirable sign, symptom or medical condition that occurred after starting study drug even if the event was not considered to be related to study drug. Percentage of participants with any AE were categorized by pasireotide incident dose classes, which were defined by total daily doses ranges (<1200 μg/d, 1200 to <1500 μg/d, ≥ 1500 μg/d).
Time Frame: From start of study drug treatment up to end of study (approximately 111 months)
Population: Safety population included all participants who had received pasireotide s.c. in the extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Pasireotide s.c. <1200 μg/d | Pasireotide s.c. 1200 to <1500 μg/d | Pasireotide s.c. ≥1500 μg/d
Number analyzed (Participants) | 30 | 30 | 12
percentage of participants | 80.0 | 86.7 | 91.7

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were monitored from date of First Participant First Visit (FPFV) until Last Participant Last Visit (LPLV). All other adverse events are monitored from First Participant First Treatment until Last Participant Last Visit (approximately 111 months).
Arm/Group | Pasireotide s.c. <1200 μg/d | Pasireotide s.c. 1200 to <1500 μg/d | Pasireotide s.c. ≥1500 μg/d
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/30 | 4/30 | 2/12
Other Adverse Events (participants affected / at risk) | 21/30 | 25/30 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide s.c. <1200 μg/d (N=30) | Pasireotide s.c. 1200 to <1500 μg/d (N=30) | Pasireotide s.c. ≥1500 μg/d (N=12)
Acromegaly (Endocrine disorders) | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide s.c. <1200 μg/d (N=30) | Pasireotide s.c. 1200 to <1500 μg/d (N=30) | Pasireotide s.c. ≥1500 μg/d (N=12)
Hypertension (Vascular disorders) | 2 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 1
Chest pain (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 4 | 1
Paraesthesia (Nervous system disorders) | 2 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 4 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 10 | 1
Oesophageal spasm (Gastrointestinal disorders) | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Burn infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 2
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 3 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.